CLINICAL TRIAL: NCT05336890
Title: Post-Vent, the Sequelae: Personalized Prognostic Modeling for Consequences of Neonatal Intermittent Hypoxemia in Preterm Infants at Pre-School Age
Status: Recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: University of Virginia (Other); Case Western Reserve University (Other); University of Miami (Other); Northwestern University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: HSR210359; 1R01HL157256-01A1 (NIH)
Record Dates: First submitted 2022-04-14; First posted 2022-04-20 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Premature Birth; Asthma in Children; Sleep-Disordered Breathing; Neurodevelopmental Disorders
MeSH Terms: conditions — Premature Birth; Sleep Apnea Syndromes; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite improved survival of extremely premature infants in recent decades, neonatal intensive care unit (NICU) graduates are diagnosed with asthma, sleep disordered breathing (SDB) in childhood, and neurodevelopmental impairments (NDI) at significant rates, disproportionate to their term peers. Early detection and intervention are critical to mitigate the impact of these impairments. Mechanisms leading from premature birth to these undesirable outcomes remain unclear, and accurate prognostic measures are lacking.

This study wants to learn if these problems are related to certain patterns of breathing that babies had while they were in the NICU.

DETAILED DESCRIPTION:
Asthma, SDB, and NDI are common consequences of preterm birth with significant impact on child and family quality of life and public health. To date, the mechanisms leading to these outcomes remain unclear, and improvements in neonatal care have not improved these outcomes. While early detection and intervention can reduce the burden of these outcomes, methods for early identification of infants destined for these morbidities is currently lacking. Utilizing the Pre-Vent cohort to investigate potential underlying causes and identify predictors for these conditions as we propose here is essential to inform future prevention and intervention strategies that promote optimal health and development.

Recent compelling data indicate that early postnatal intermittent hypoxemia (IH) events may play a role in undesirable outcomes. Early postnatal IH events in extremely preterm infants are associated with bronchopulmonary dysplasia (BPD), asthma medication at 2 years, and NDI at 18 months. The ability of IH to perturb maturation of long-term respiratory control has been demonstrated in neonatal rodents consistent with preterm infants being at heightened risk for childhood SDB. Although evidence is emerging that IH events are linked to poor outcomes in premature infants, the specific relationship between distinct IH patterns (e.g. duration, timing, frequency, and nadir) and longer-term respiratory and neurologic function remains to be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in any Institutional Review Board (IRB) protocol of the Pre-Vent Study that had signed consent, or in any IRB protocol of the Pre-Vent Study that authorized re-contact for future research
* Born <29 weeks gestational age
* Age at enrollment less than 7 years old

Exclusion Criteria:

* Subject was withdrawn from the Pre-Vent study after signing Pre-Vent consent form, for any reason
* Subject had no physiological data recorded as part of Pre-Vent
* Lack of regulatory approval from local IRB or Department of Children and Family Services (DCFS) to recontact subjects
* Adopted by non-consenting family
* Parent refused further contact, prior to approach for Post-Vent
* Infant enrolled in Pre-Vent at Washington University St Louis, which is not a Post-Vent participating site.

Ages: 30 Weeks to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will be drawn from surviving, previously consented children in the existing Pre-Vent study cohort or in any IRB protocol of the Pre-Vent study that authorized re-contact for future research, which was drawn from Neonatal Intensive Care Unit Populations in Chicago, IL; Cleveland, OH; Birmingham, AB; or Miami, FL, USA.
  Up to 500 children will be enrolled after parent/guardian provides informed consent.
  Parents, guardians or primary caretakers will act as proxies for providing information about the children.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Asthma | 5 years ± 6 months of age
  Doctor diagnosed asthma as assessed in the International Study on Asthma and Allergies in Childhood questionnaire (ISAAC)
Sleep Disordered Breathing (SDB) | 5 years ± 6 months of age
  Sleep-Related Breathing Disorder (SRBD) score >= 0.33. Scores >0.33 are considered positive and suggestive of high-risk for a pediatric sleep-related breathing disorder.
Neurodevelopmental Impairment (NDI) | 5 years ± 6 months of age
  ≤10th percentile in any of the National Institutes of Health (NIH) Toolbox domains may indicate neurodevelopmental impairment.

SECONDARY OUTCOMES:
Respiratory Symptoms | 5 yr. (+/- 6 months)
  Respiratory Symptoms reported on the ISAAC Questionnaire
Medically attended respiratory illnesses | 5 yr. (+/- 6 months)
  Medically attended respiratory illnesses in the past year by ISAAC questionnaire
Asthma Severity | 5 yr. (+/- 6 months)
  Asthma Severity by Modified Composite Asthma Severity Score (MCASI). Minimum value = 0. Max value = 21. Higher scores mean a worse outcome.
Sleep Disordered Breathing (SDB) | 5 yr. (+/- 6 months)
  Score on SDB questionnaire. Scores >0.33 are considered positive and suggestive of high-risk for a pediatric sleep-related breathing disorder.
Motor Function | 5 yr. (+/- 6 months)
  Motor Function based on NIH Toolbox Motor Battery
Gross Motor Function | 5 yr. (+/- 6 months)
  Motor Function based on Gross Motor Functional Classification System
Cognitive Function | 5 yr. (+/- 6 months)
  Cognitive Function based on NIH Toolbox Cognitive Battery
Executive Function | 5 yr. (+/- 6 months)
  Executive Function based on Behavior rating inventory of executive function
Social, Emotional and Behavioral Outcomes | 5 yr. (+/- 6 months)
  Social, Emotional and Behavioral Outcomes based on NIH Toolbox Parent Proxy Emotion Battery
Sensory Outcomes: Odor Identification | 5 yr. (+/- 6 months)
  Sensory Outcomes based on NIH Toolbox Odor Identification Test
Sensory Outcomes: Acuity | 5 yr. (+/- 6 months)
  Sensory Outcomes based on NIH Toolbox Visual Acuity Test
Pediatric Quality of life | 5 yr. (+/- 6 months)
  Quality of life as assessed by the Pediatric Quality of Life parent proxy questionnaire
Health utilization | 5 yr. (+/- 6 months)
  Health utilization, based on broad health parent questionnaire
Medications | 5 yr. (+/- 6 months)
  Medications based on broad health parent questionnaire
Doctor Diagnosed Asthma | 6 mo through 5 yr. +6 months
  Doctor Diagnosed Asthma based on ISAAC
Respiratory Symptoms | 6 mo through 5 yr. +6 months
  Respiratory Symptoms based on ISAAC
Medically attended respiratory illnesses | 6 mo through 5 yr. +6 months
  Medically attended respiratory illnesses in past year based on broad health parent questionnaire
Asthma Severity: Modified Composite Asthma Severity Index(MCASI) | 6 mo through 5 yr. +6 months
  Asthma Severity by MCASI score. Minimum value = 0. Max value = 21. Higher scores mean a worse outcome.
Asthma Severity: Global Initiative for Asthma criteria (GINA) | 6 mo through 5 yr. +6 months
  Asthma Severity using GINA criteria based on broad health parent questionnaire. A score of 19 or less indicates poorly controlled asthma, while a score greater than 19 indicates well-controlled asthma.
Health utilization | 6 mo through 5 yr. +6 months
  Health utilization, based on parent broad health questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Debra Weese-Mayer, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Anna Maria Hibbs, MD, Principal Investigator — Case Western Reserve University; Ambalavanan Namasivayam, MD, Principal Investigator — University of Alabama at Birmingham; Nelson Claure, MSc, PhD, Principal Investigator — University of Miami; Randall Moorman, MD, Principal Investigator — University of Virginia
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No